CLINICAL TRIAL: NCT01949480
Title: Comparison Of Ultrasound-Assisted Paravertebral Block And Traditional Paravertebral Block For Pain Control After Thoracic Surgery, A Prospective Randomized Trial
Brief Title: Ultrasound-Assisted Paravertebral Block v. Traditional Paravertebral Block For Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Anna Uskova, Clinical Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO09090367
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-08

CONDITIONS: Paravertebral Peripheral Nerve Block; Acute Pain Management
Keywords: Peripheral nerve block; Ultrasound guidance; Postoperative pain management post status thoracotomy; Postoperative pain management post status VATS
MeSH Terms: interventions — Thoracotomy; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional approach paravertebral nerve block (Active Comparator): After final needle placement, a hanging drop technique will be used to rule out intrapleural placement while the patient inhales and exhales deeply. After correct needle placement, 10 mL of 0.5% Ropivacaine will be injected incrementally through each needle after negative aspiration, followed by insertion of the nerve block catheter to a depth 5 cm beyond the tip of the needle. An additional 10 mL of 0.5% Ropivacaine will then be injected in 5 mL increments with negative aspiration in between, through the catheter yielding a total activation dose of 20 ml of 0.5% Ropivacaine. The catheter will be secured with Steri-strips and a transparent occlusive dressing.
  Interventions: Procedure: Thoracotomy; Procedure: Video-Assisted Thoracoscopic Surgery (VATS)
- Ultrasound assisted paravertebral nerve block (Experimental): The 22 gauge catheter will be threaded through the needle and placed at previously found distance to paravertebral space on obtained ultrasound image. An additional 10 ml of 0.5% Ropivacaine will be administered through the catheter yielding a total activation dose of 20 ml of 0.5% Ropivacaine. The catheter will be secured with Steri-strips and a transparent occlusive dressing.
  Interventions: Procedure: Thoracotomy; Procedure: Video-Assisted Thoracoscopic Surgery (VATS)

INTERVENTIONS:
Procedure: Thoracotomy
Procedure: Video-Assisted Thoracoscopic Surgery (VATS)

SUMMARY:
The overall purpose of this research study is to compare the effectiveness of ultrasound assisted paravertebral block placement versus traditional "blind" technique for postoperative analgesia following thoracotomy or visually assisted thoracoscopic surgery.

DETAILED DESCRIPTION:
The purpose of this project is to determine if there is a difference between paravertebral block performed with ultrasound assistance and paravertebral block performed with traditional technique in terms of twenty - four hour hydromorphone (dilaudid) consumption and visual analogue pain scores at rest or with deep breathing at twenty - four hours. This study will determine if ultrasound technique used for placement of paravertebral catheter facilitates safety of paravertebral catheterization and improves therapeutic effect of paravertebral blockade for pain control after thoracotomy. The investigators will also examine if ultrasound assisted paravertebral blockade improves pulmonary status in post-thoracotomy patient.

ELIGIBILITY:
Inclusion Criteria:

* 1. American Society of Anesthesiologists (ASA) I-III subjects
* 2. Ages 18-75 years
* 3. BMI < 40
* 4. Scheduled for elective thoracic surgery at University of Pittsburgh Medical Center (UPMC) Passavant and Shadyside Hospitals in Pittsburgh, Pennsylvania
* 5. Patients willing and able to provide informed consent

Exclusion Criteria:

* 1) Age younger than 18 years or older than 75 years
* (2) Any contraindication to the placement of unilateral thoracic paravertebral catheter, including local infection, hypocoagulable state.
* (3) American Society of Anesthesiologists physical status IV or greater
* (4) chronic painful conditions
* (5) preoperative opioid use
* (6) coagulation abnormalities or patients who are expected to be on therapeutic anticoagulants postoperatively
* (7) allergy to lidocaine, ropivacaine or bupivacaine
* (8) personal or family history of malignant hyperthermia
* (9) serum creatinine greater than 1.4 g/dl
* (10) pregnancy or lactating.The pregnancy status will be determined by history and prior pregnancy testing when appropriate
* (11) having an altered mental status (not oriented to place, person, or time) or emergency surgery
* (12) comorbid conditions such as sepsis, unstable angina, congestive heart failure, moderate to severe valvular heart disease, severe chronic obstructive pulmonary disease (COPD)
* (13) patient's inability to provide adequate informed consent
* (14) patient refusal to nerve blocks and/or participation in the study
* (15) respiratory support via ventilator post
* (16) non English speaking
* (17) allergy to contrast of iodine
* (18) emergency surgery or any other non-elective procedure
* (19) unstable vertebral and transverse process fractures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2014-06-05 (Actual); Study Completion 2014-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Uskova, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania
  - UPMC Passavant, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Richardson J, Sabanathan S, Jones J, Shah RD, Cheema S, Mearns AJ. A prospective, randomized comparison of preoperative and continuous balanced epidural or paravertebral bupivacaine on post-thoracotomy pain, pulmonary function and stress responses. Br J Anaesth. 1999 Sep;83(3):387-92. doi: 10.1093/bja/83.3.387. PMID 10655907
- [Background] Perttunen K, Nilsson E, Heinonen J, Hirvisalo EL, Salo JA, Kalso E. Extradural, paravertebral and intercostal nerve blocks for post-thoracotomy pain. Br J Anaesth. 1995 Nov;75(5):541-7. doi: 10.1093/bja/75.5.541. PMID 7577277
- [Background] Matthews PJ, Govenden V. Comparison of continuous paravertebral and extradural infusions of bupivacaine for pain relief after thoracotomy. Br J Anaesth. 1989 Feb;62(2):204-5. doi: 10.1093/bja/62.2.204. PMID 2923769
- [Background] Lonnqvist PA, MacKenzie J, Soni AK, Conacher ID. Paravertebral blockade. Failure rate and complications. Anaesthesia. 1995 Sep;50(9):813-5. doi: 10.1111/j.1365-2044.1995.tb06148.x. PMID 7573876
- [Background] Vogt A, Stieger DS, Theurillat C, Curatolo M. Single-injection thoracic paravertebral block for postoperative pain treatment after thoracoscopic surgery. Br J Anaesth. 2005 Dec;95(6):816-21. doi: 10.1093/bja/aei250. Epub 2005 Sep 30. PMID 16199417
- [Background] Ganapathy S, Murkin JM, Boyd DW, Dobkowski W, Morgan J. Continuous percutaneous paravertebral block for minimally invasive cardiac surgery. J Cardiothorac Vasc Anesth. 1999 Oct;13(5):594-6. doi: 10.1016/s1053-0770(99)90015-0. No abstract available. PMID 10527232
- [Background] Weltz CR, Greengrass RA, Lyerly HK. Ambulatory surgical management of breast carcinoma using paravertebral block. Ann Surg. 1995 Jul;222(1):19-26. doi: 10.1097/00000658-199507000-00004. PMID 7618963
- [Background] Klein SM, Bergh A, Steele SM, Georgiade GS, Greengrass RA. Thoracic paravertebral block for breast surgery. Anesth Analg. 2000 Jun;90(6):1402-5. doi: 10.1097/00000539-200006000-00026. PMID 10825328
- [Background] Pusch F, Freitag H, Weinstabl C, Obwegeser R, Huber E, Wildling E. Single-injection paravertebral block compared to general anaesthesia in breast surgery. Acta Anaesthesiol Scand. 1999 Aug;43(7):770-4. doi: 10.1034/j.1399-6576.1999.430714.x. PMID 10456819
- [Background] Richardson J, Vowden P, Sabanathan S. Bilateral paravertebral analgesia for major abdominal vascular surgery: a preliminary report. Anaesthesia. 1995 Nov;50(11):995-8. doi: 10.1111/j.1365-2044.1995.tb05939.x. PMID 8678263
- [Background] Kirvela O, Antila H. Thoracic paravertebral block in chronic postoperative pain. Reg Anesth. 1992 Nov-Dec;17(6):348-50. PMID 1286056
- [Background] Karmakar MK, Chui PT, Joynt GM, Ho AM. Thoracic paravertebral block for management of pain associated with multiple fractured ribs in patients with concomitant lumbar spinal trauma. Reg Anesth Pain Med. 2001 Mar-Apr;26(2):169-73. doi: 10.1053/rapm.2001.21086. PMID 11251143
- [Background] Chelly JE. Peripheral Nerve Blocks: A Color Atlas. 2009. Third Edition. Lippincott Williams and Wilkins.
- [Background] Terheggen MA, Wille F, Borel Rinkes IH, Ionescu TI, Knape JT. Paravertebral blockade for minor breast surgery. Anesth Analg. 2002 Feb;94(2):355-9, table of contents. doi: 10.1097/00000539-200202000-00023. PMID 11812698
- [Background] Evans PJ, Lloyd JW, Wood GJ. Accidental intrathecal injection of bupivacaine and dextran. Anaesthesia. 1981 Jul;36(7):685-7. doi: 10.1111/j.1365-2044.1981.tb08781.x. PMID 6168207
- [Background] Chan VWS, Perlas A, Rawson R, Odukoya O. Ultrasound-guided supraclavicular brachial plexus block. Anesth Analg. 2003 Nov;97(5):1514-1517. doi: 10.1213/01.ANE.0000062519.61520.14. PMID 14570677
- [Background] Marhofer P, Sitzwohl C, Greher M, Kapral S. Ultrasound guidance for infraclavicular brachial plexus anaesthesia in children. Anaesthesia. 2004 Jul;59(7):642-6. doi: 10.1111/j.1365-2044.2004.03669.x. PMID 15200537
- [Background] Luyet C, Eichenberger U, Greif R, Vogt A, Szucs Farkas Z, Moriggl B. Ultrasound-guided paravertebral puncture and placement of catheters in human cadavers: an imaging study. Br J Anaesth. 2009 Apr;102(4):534-9. doi: 10.1093/bja/aep015. Epub 2009 Feb 24. PMID 19244265
- See also: University of Pittsburgh Institutional Review Board — http://www.irb.pitt.edu/
- See also: University of Pittsburgh Department of Anesthesiology — http://www.anes.upmc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 1, 2013- May 29 2014, 45 patients scheduled for thoracic surgery were approached in the preoperative setting and consented for the study.
Pre-assignment Details: 3 of the 45 consented patients were excluded because they did not meet inclusion criteria
Groups:
- Traditional Approach Paravertebral Nerve Block: After final needle placement, a hanging drop technique will be used to rule out intrapleural placement while the patient inhales and exhales deeply. After correct needle placement, 10 mL of 0.5% Ropivacaine will be injected incrementally through each needle after negative aspiration, followed by insertion of the nerve block catheter to a depth 5 cm beyond the tip of the needle. An additional 10 mL of 0.5% Ropivacaine will then be injected in 5 mL increments with negative aspiration in between, through the catheter yielding a total activation dose of 20 ml of 0.5% Ropivacaine. The catheter will be secured with Steri-strips and a transparent occlusive dressing.
  Thoracotomy
  Video-Assisted Thoracoscopic Surgery (VATS)
- Ultrasound Assisted Paravertebral Nerve Block: The 22 gauge catheter will be threaded through the needle and placed at previously found distance to paravertebral space on obtained ultrasound image. An additional 10 ml of 0.5% Ropivacaine will be administered through the catheter yielding a total activation dose of 20 ml of 0.5% Ropivacaine. The catheter will be secured with Steri-strips and a transparent occlusive dressing.
  Thoracotomy
  Video-Assisted Thoracoscopic Surgery (VATS)
Period: Overall Study
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Started | 20 | 22
Completed | 15 | 14
Not Completed | 5 | 8
Not completed — Physician Decision | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 12 | 11 | 23
Age, Continuous [Mean (Full Range); unit: years] | 68 [59.5 to 71.5] | 64 [57 to 70] | 66 [57 to 71.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption at 24 Hours Postoperatively
Description: Hydromorphone (Dilaudid) consumption or opiate equivalent at 24-hour interval post PCA initiation at the post-anesthesia care unit (PACU).
Time Frame: 24 hours after patient-controlled analgesia (PCA) was initiated
Population: There are only 13 participants in the Ultrasound Assisted paravertebral nerve block arm, because (n=1) 1 participant was excluded from analysis due to shoulder dislocation during surgical positioning.
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 13
mg | 5.75 [3.9 to 7.59] | 6.38 [4.09 to 8.66]
Statistical Analysis 1: Comparison: Traditional Approach Paravertebral Nerve Block vs Ultrasound Assisted Paravertebral Nerve Block; Test type: Non-Inferiority — To detect an effect size of 0.92 SD units with a power of 81% and alpha level of 0.05, a total sample size of 40 patients (20 patients/group) was calculated; p = 0.643, t-test, 2 sided

2. Secondary Outcome: Sensory Level
Description: Sensory level as assessed by temperature and pin prick test assessed every 5 min for 30 min after nerve block as defined as the patient returning to their bed. Data below are in number of patients who didn't have any change during the ice and pin prik test.
Time Frame: 6 assessments starting 5 minutes after nerve block and ending 30 minutes after nerve block.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 13
Participants | 3 | 1

3. Secondary Outcome: Pain 11-point Numerical Rating Scale (NRS)at Rest and With Deep Breathing
Description: The pain level assessed using an 11-point numerical rating scale (NRS) with 0 indicating no pain and 10 indicating the worst pain possible with deep breathing and rest at 24 hours post PCA initiation.
Time Frame: 24 hours post PCA initiation
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 13
units on a scale
  NRS at rest after 24 hrs | 1.73 [1.04 to 2.43] | 2.92 [1.99 to 3.86]
  NRS during deep inspiration at 24 hrs | 4 [2.58 to 5.42] | 4.77 [3.56 to 5.98]
Statistical Analysis 1: Comparison: Traditional Approach Paravertebral Nerve Block vs Ultrasound Assisted Paravertebral Nerve Block; This p-value is calculated for the NRS at rest; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = .077, t-test, 2 sided
Statistical Analysis 2: Comparison: Traditional Approach Paravertebral Nerve Block vs Ultrasound Assisted Paravertebral Nerve Block; This p-value is calculated for the NRS during deep inspiration at 24 hrs; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.39, t-test, 2 sided

4. Secondary Outcome: Number of Local Anesthetic Boluses Requested by PCA
Description: The number of local anesthetic boluses over 24- hour period post PCA initiation will also be recorded.
Time Frame: 24 hours postoperatively
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Number of boluses requested
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 13
Number of boluses requested | 27.5 [13.5 to 57.2] | 48 [17 to 63]
Statistical Analysis 1: Comparison: Traditional Approach Paravertebral Nerve Block vs Ultrasound Assisted Paravertebral Nerve Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.605, t-test, 2 sided

5. Secondary Outcome: Total Local Anesthetic Infusions Over 24- Hour Period
Description: The total local anesthetic infusions over 24- hour period.
Time Frame: 24 hours postoperatively
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 13
mL | 173 [168 to 184] | 186 [175 to 197]
Statistical Analysis 1: Comparison: Traditional Approach Paravertebral Nerve Block vs Ultrasound Assisted Paravertebral Nerve Block; This p-value is for the Local Anesthetic infused in 24 hrs; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.104, t-test, 2 sided

6. Secondary Outcome: Inspired Oxygen Concentration and Blood Oxygen Saturation (SpO2)
Description: Inspired oxygen concentration and SpO2 preoperatively and at 24 - hour interval. Value reported is an average of the preoperative and the 24-hour postoperative SpO2 measurements.
Time Frame: Pre-operatively and at 24 hour post-operative
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage of SpO2
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 13
Percentage of SpO2 | 95 [94 to 96] | 94 [93 to 95]
Statistical Analysis 1: Comparison: Traditional Approach Paravertebral Nerve Block vs Ultrasound Assisted Paravertebral Nerve Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.308, t-test, 2 sided

7. Secondary Outcome: Incentive Spirometry
Description: Inspiratory Volume as measured by incentive spirometer preoperatively and at 24 hours post PCA initiation. The data is reported as a percentage in change from per-surgery measurements (post-surgery/pre-surgery).
Time Frame: Preoperatively and Postoperatively
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage in change from per-surgery
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 13
percentage in change from per-surgery | 0.658 [0.544 to 0.773] | 0.716 [0.575 to 0.857]
Statistical Analysis 1: Comparison: Traditional Approach Paravertebral Nerve Block vs Ultrasound Assisted Paravertebral Nerve Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.487, t-test, 2 sided

8. Secondary Outcome: Respiratory Rate
Description: Respiratory rate (RR) per minute after surgery.
Time Frame: 24 hours postoperatively
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: breaths per one minute
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 13
breaths per one minute | 17 [15.8 to 18.2] | 17.7 [15.9 to 19.5]
Statistical Analysis 1: Comparison: Traditional Approach Paravertebral Nerve Block vs Ultrasound Assisted Paravertebral Nerve Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.493, t-test, 2 sided

9. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Forced vital capacity (FVC) measured preoperatively and at 24 - hour interval. Then values were analyzed as percentage in change from per-surgery measurement (post-surgery/pre-surgery).
Time Frame: Preoperatively and postoperatively
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage in change from per-surgery
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 13
percentage in change from per-surgery | 0.551 [0.403 to 0.699] | 0.504 [0.395 to 0.613]
Statistical Analysis 1: Comparison: Traditional Approach Paravertebral Nerve Block vs Ultrasound Assisted Paravertebral Nerve Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.574, t-test, 2 sided

10. Secondary Outcome: Forced Expiratory Volume in 1 Sec (FEV1)
Description: Forced expiratory volume in 1 sec (FEV1) preoperatively and at 24 - hour interval. Then the values were analyzed as percentage in change from per-surgery measurement (post-surgery/pre-surgery).
Time Frame: Preoperatively and postoperatively
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage in change from per-surgery
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 13
percentage in change from per-surgery | 0.561 [0.4 to 0.722] | 0.571 [0.466 to 0.675]
Statistical Analysis 1: Comparison: Traditional Approach Paravertebral Nerve Block vs Ultrasound Assisted Paravertebral Nerve Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.913, t-test, 2 sided

11. Secondary Outcome: Peak Expiratory Flow Rate(PEF)
Description: Peak expiratory flow rate preoperatively (PEF) and at 24 - hour interval. Then values were analyzed as percentage in change from per-surgery measurement (post-surgery/pre-surgery).
Time Frame: Preoperatively and postoperatively
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage in change from per-surgery
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 13
percentage in change from per-surgery | 0.568 [0.4 to 0.735] | 0.542 [0.42 to 0.664]
Statistical Analysis 1: Comparison: Traditional Approach Paravertebral Nerve Block vs Ultrasound Assisted Paravertebral Nerve Block; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.783, t-test, 2 sided

12. Secondary Outcome: Total Number of Local Anesthetic Boluses in 24 Hours
Description: Total Number of Local Anesthetic bolus doses given within the 24-hours post-operatively.
Time Frame: postoperatively, up to 24 hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of boluses
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
Number analyzed (Participants) | 15 | 13
number of boluses | 1 [0 to 1.5] | 2 [1 to 4]

ADVERSE EVENTS:
Time Frame: Adverse events collected for 24 hours post-operatively
Description: If the adverse event (AE) resulted in prolonged hospitalization, serious illness or death, it would be considered a Serious Adverse Event (SAE).
Arm/Group | Traditional Approach Paravertebral Nerve Block | Ultrasound Assisted Paravertebral Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 2/20 | 3/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Approach Paravertebral Nerve Block (N=20) | Ultrasound Assisted Paravertebral Nerve Block (N=22)
Catheter leaking (Surgical and medical procedures) | 2 (2) | 3 (3) — Catheter leaking/repositioned in pleural space

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes